CLINICAL TRIAL: NCT04626297
Title: A Phase 3, 16-week, Randomized, Double-Blind, Placebo-Controlled, Parallel- Group Study to Assess the Impact of Lebrikizumab on Vaccine Responses in Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Lebrikizumab (LY3650150) on Vaccine Response in Adults With Atopic Dermatitis (ADopt-VA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17946; J2T-MC-KGAK (Other: Eli Lilly and Company); 2020-002572-12 (EudraCT Number)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lebrikizumab (Experimental): Participants received a loading dose of 500 milligram (mg) lebrikizumab injection administered subcutaneously (SC) at baseline and week 2, and 250 mg once every two weeks (Q2W) from week 4 to 14.
  Interventions: Drug: Lebrikizumab
- Placebo (Placebo Comparator): Participants received placebo SC injection Q2W from baseline to week 14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Given SC
  Other Names: LY3650150; DRM06
  Arms: Lebrikizumab
Drug: Placebo — Given SC
  Arms: Placebo

SUMMARY:
The reason for this study is to assess the impact of lebrikizumab on vaccine immune response in adult participants with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic atopic dermatitis (AD) according to American Academy of Dermatology Consensus Criteria that has been present for ≥1 year before screening.
* Eczema Area and Severity Index (EASI) score ≥16 at the baseline visit.
* Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the baseline visit.
* ≥10% Body Surface Area (BSA) of AD involvement at the baseline visit.
* History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.
* Have not received any tetanus-containing vaccine within approximately 5 years of baseline.
* Have never received a meningococcal conjugate vaccine or have received not more than 1 prior MCV dose at least 4 years prior to baseline, of a vaccine containing 1 or more meningococcal serogroups (serogroups A, C, W, Y).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * a. Female participants of childbearing potential: must agree to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method during the treatment period and for at least 18 weeks after the last dose of study drug. Women of non-childbearing potential (non-WOCBP) may participate without any contraception requirements.
  * b. Male participants are not required to use any contraception except in compliance with specific local government study requirements.

Exclusion Criteria:

* Recurring herpes simplex, herpes zoster, recurring cellulitis, chronic osteomyelitis
* Evidence of active or chronic hepatitis
* History of human immunodeficiency virus (HIV) infection or positive HIV serology.
* Presence of skin comorbidities that may interfere with study assessments.
* History of malignancy, including mycosis fungoides, within 5 years before screening, except completely treated in situ carcinoma of the cervix or completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
* Uncontrolled chronic disease that might require bursts of oral corticosteroids, e.g., co-morbid severe uncontrolled asthma.
* Have a prior history of Guillain-Barre syndrome.
* Allergic to latex.
* History of past vaccination allergy or Arthus-type hypersensitivity.
* Have an uncontrolled seizure disorder.
* Have known hypogammaglobulinemia or a screening serum immunoglobulin G (IgG) or immunoglobulin A (IgA) concentration less than the lower limit of the reporting laboratory's reference range.
* Treated with topical corticosteroids (TCS), calcineurin inhibitors, or phosphodiesterase-4 inhibitors such as crisaborole within 1 week prior to the baseline visit.
* Treated with the following prior to baseline visit:

  * a. An investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer
  * b. B Cell-depleting biologics, including rituximab, within 6 months
  * c. Other biologics within 5 half-lives (if known) or 8 weeks, whichever is longer
* Received a Bacillus Calmette-Guerin (BCG) vaccination or treatment within 12 months of screening, or treated with a live (attenuated) vaccine within 12 weeks of the baseline visit or planned during the study.
* A contraindication to the Tdap vaccine or mean corpuscular volume (MCV).
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (85):
- United States (85):
  - Clinical Research Center of Alabama- Birmingham, Birmingham, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Wallace Medical Group, Inc., Beverly Hills, California
  - First OC Dermatology, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Axon Clinical Research, Inglewood, California
  - Sunwise Clinical Research, Lafayette, California
  - Avance Trials, Laguna Niguel, California
  - Keck School of Medicine University of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - LA Universal Research Center, INC, Los Angeles, California
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Dermatology Clinical Trials, Newport Beach, California
  - Cura Clinical Research, Palmdale, California
  - MD Strategies Research Centers MDSRC, San Diego, California
  - University Clinical Trials, San Diego, California
  - Synergy Dermatology, San Francisco, California
  - Care Access Research, San Jose, California
  - San Luis Dermatology & Laser Clinic, San Luis Obispo, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - C&R Research Services USA, Kendall, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Sanchez Clinical Research Inc, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Florida Research Center, Inc, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - Tampa General Hospital, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - Georgia Skin & Cancer Clinic, Savannah, Georgia
  - Sneeze, Wheeze, & Itch Associates LLC, Normal, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Kansas Medical Clinic, an Elligo Health Research, Inc., Shawnee Mission, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Tulane Univ School of Med, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Oakland Dermatology, Auburn Hills, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Advanced Dermatology of the Midlands, Omaha, Nebraska
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Skin Laser and Surgery Specialists, a Division of Schweiger Dermatology, Hackensack, New Jersey
  - JUVA Skin & Laser Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Central States Research, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Peak Research LLC, Upper Saint Clair, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Arlington Research Center, Inc, Arlington, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Modern Research Associates, Dallas, Texas
  - Austin Institute for Clinical Research, Dripping Springs, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Laredo Dermatology Associates P.A., Laredo, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Velocity Clinical Research - Woseth Dermatology, Salt Lake City, Utah
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Soung J, Laquer V, Merola JF, Moore A, Elmaraghy H, Hu C, Piruzeli MLB, Pierce E, Garcia Gil E, Jarell AD. The Impact of Lebrikizumab on Vaccine-Induced Immune Responses: Results from a Phase 3 Study in Adult Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Aug;14(8):2181-2193. doi: 10.1007/s13555-024-01217-w. Epub 2024 Jul 15. PMID 39009804
- See also: A Study of Lebrikizumab (LY3650150) on Vaccine Response in Adults With Atopic Dermatitis (ADopt-VA) — https://trials.lillytrialguide.com/en-US/trial/589axvNecFXMpOxA4PGIx3

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo subcutaneous (SC) injection once every two weeks (Q2W) from baseline to week 14.
- Lebrikizumab 250 mg: Participants received a loading dose of 500 milligram (mg) lebrikizumab injection administered SC at baseline and week 2, and 250 mg Q2W from week 4 to 14.
Period: Overall Study
Arm/Group | Placebo | Lebrikizumab 250 mg
Started | 127 | 127
Received at Least 1 Dose of Study Drug | 127 | 127
Completed | 88 | 113
Not Completed | 39 | 14
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 7 | 3
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 20 | 6
Not completed — Sponsor decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Lebrikizumab 250 mg: Participants received a loading dose of 500 mg lebrikizumab injection administered SC at baseline and week 2, and 250 mg Q2W from week 4 to 14.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lebrikizumab 250 mg | Total
Number analyzed (Participants) | 127 | 127 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (10.14) | 35.2 (11.54) | 35.6 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 139
  Male | 60 | 55 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 49 | 94
  Not Hispanic or Latino | 82 | 77 | 159
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 18 | 16 | 34
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 29 | 29 | 58
  White | 72 | 74 | 146
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127 | 127 | 254

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Develop a Booster Response to Tetanus Toxoid 4 Weeks After Tdap (Tetanus-diphtheria-pertussis) Vaccine Administration
Description: Booster response to tetanus toxoid is defined as: ≥4-fold increase in anti-tetanus toxoid immunoglobulin G (IgG) antibody concentration if the pre-vaccination level was >0.10 International units per milliliter (IU/mL) and ≤2.7 IU/mL; OR ≥2-fold increase in anti-tetanus toxoid IgG antibody concentration if the pre-vaccination level was >2.7 IU/mL; OR ≥4-fold increase in anti-tetanus toxoid IgG antibody concentration and a post-vaccination level ≥0.10 IU/mL if the pre-vaccination level was ≤0.10 IU/mL
Time Frame: Week 16
Population: All randomized participants who received at least 1 dose of study drug, had no significant protocol deviations, and had non-missing sero-response data to Tdap vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 79 | 106
percentage of participants | 73.4 | 73.6
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; Risk Difference (RD) = 0.3, 90% CI 2-sided [-10.2 to 11.2]

2. Primary Outcome: Percentage of Participants Who Have Positive Antibody Response to Meningococcus C Antigen 4 Weeks After Meningococcal Conjugate Vaccine (MCV) Administration
Description: Positive antibody response to Meningococcus C antigen as measured by group C serum bactericidal antibodies is defined as: post-vaccination rabbit complement serum bactericidal assay (rSBA) titer ≥4 times the lower limit of quantitation (LLOQ), if the pre-vaccination rSBA titer is less than the LLOQ; OR post-vaccination rSBA titer ≥4 times the pre-vaccination titer, if the pre-vaccination rSBA titer is greater than or equal to the LLOQ.
Time Frame: Week 16
Population: All randomized participants who received at least 1 dose of study drug, had no significant protocol deviations, and had non-missing sero-response data to MCV.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 80 | 99
percentage of participants | 75 | 86.9
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; Risk Difference (RD) = 12.2, 90% CI 2-sided [2.5 to 22.0]

3. Secondary Outcome: Percentage of Participants Achieving an Investigator Global Assessment (IGA) Score of 0 or 1 and a Reduction of ≥2 Points From Baseline
Description: The IGA measures the investigator's global assessment of the participants overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. Markov Chain Monte Carlo Multiple Imputation (MCMC-MI) was used to handle missing data.
Time Frame: Week 16
Population: All randomized participants. Following a site audit and findings of non-compliance, two investigational sites with seven participants were excluded from the analysis as the data was considered unreliable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 122 | 125
percentage of participants | 18.9 [11.4 to 26.3] | 40.6 [31.8 to 49.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.7, 95% CI 2-sided [10.3 to 33.2]

4. Secondary Outcome: Percentage of Participants Achieving a ≥75% Reduction From Baseline in Eczema Area and Severity Index Score (EASI-75)
Description: The EASI-75 is defined as a ≥ 75% improvement from baseline in the EASI score. EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs, by scoring the extent of disease (percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed. The final EASI score will be obtained by weight-averaging these 4 scores and will range from 0 to 72. A higher score represents greater disease severity. MCMC-MI was used to handle missing data.
Time Frame: Week 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 122 | 125
percentage of participants | 32.7 [23.5 to 41.9] | 58.0 [49.1 to 66.9]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.3, 95% CI 2-sided [12.6 to 38]

5. Secondary Outcome: Percentage of Participants Achieving ≥90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI-90)
Description: The EASI-90 is defined as a ≥ 90% improvement from baseline in the EASI score. EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs, by scoring the extent of disease (percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed. The final EASI score will be obtained by weight-averaging these 4 scores and will range from 0 to 72. A higher score represents greater disease severity. MCMC-MI was used to handle missing data.
Time Frame: Week 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 122 | 125
percentage of participants | 18.9 [11.3 to 26.4] | 39.2 [30.5 to 47.9]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.3, 95% CI 2-sided [9.0 to 31.6]

6. Secondary Outcome: Percentage of Participants Achieving ≥4-Point Improvement From Baseline in Pruritus Numeric Rating Scale (NRS) Score
Description: The Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." MCMC-MI was used to handle missing data.
Time Frame: Week 16
Population: All randomized participants with a baseline pruritus NRS Score of at least 4. Following a site audit and findings of non-compliance, two investigational sites with seven participants were excluded from the analysis as the data was considered unreliable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 93 | 95
percentage of participants | 33.2 [22.6 to 43.8] | 51.7 [41.2 to 62.3]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; p = 0.138, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.9, 95% CI 2-sided [-3.8 to 27.5]

7. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA)
Description: The BSA assessment estimates the extent of disease or skin involvement with respect to AD and is expressed as a percentage of body surface area. It was assessed for 4 body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100%. BSA was calculated using the participant's palm, 1 palm = 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 for head and neck (10%), 20 for upper extremities (20%), 30 for trunk, including axilla and groin (30%), and 40 for lower extremities, including buttocks (40%). Percent of BSA for a body region = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA for an individual is arithmetic mean of % BSA of all 4 body regions and ranges from 0% to 100% with higher values representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: All randomized participants with evaluable BSA data at baseline and week 16. Following a site audit and findings of non-compliance, two investigational sites with seven participants were excluded from the analysis as the data was considered unreliable.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 85 | 110
percentage of body surface area | -19.34 (1.882) | -27.55 (1.719)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -8.21, 95% CI 2-sided [-13.04 to -3.39], Standard Error of Mean 2.447 — The mixed model repeated measures (MMRM) included treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit, geographic region, age group, baseline IGA score as fixed factors

8. Secondary Outcome: Change From Baseline in Sleep-Loss Score
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicate a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary, and the week 16 score was calculated by averaging the daily scores from the previous 7 days and the average score was used to compute a change from baseline. MCMC-MI was used to handle missing data.
Time Frame: Baseline, Week 16
Population: All randomized participants with evaluable sleep-loss score data at baseline and week 16. Following a site audit and findings of non-compliance, two investigational sites with seven participants were excluded from the analysis as the data was considered unreliable.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab 250 mg
Number analyzed (Participants) | 108 | 111
score on a scale | -0.87 (0.122) | -1.35 (0.107)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab 250 mg; Test type: Other; p = 0.001658, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.152

ADVERSE EVENTS:
Time Frame: Baseline Up To Week 26
Description: All randomized participants who received at least 1 dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | Lebrikizumab 250 mg
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127
Serious Adverse Events (participants affected / at risk) | 1/127 | 1/127
Other Adverse Events (participants affected / at risk) | 43/127 | 47/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=127) | Lebrikizumab 250 mg (N=127)
Breast cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=127) | Lebrikizumab 250 mg (N=127)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 2 (2)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site hypersensitivity (General disorders) | 0 (0) | 1 (2)
Injection site pain (General disorders) | 1 (2) | 0 (0)
Injection site pruritus (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1/67 (1) | 0/72 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3)
Covid-19 (Infections and infestations) | 5 (5) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/67 (0) | 1/72 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep inertia (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0/67 (0) | 1/72 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 (10) | 6 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04626297/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04626297/SAP_001.pdf